CLINICAL TRIAL: NCT00443859
Title: Clinical Significance of N-Terminal Pro-Brain Natriuretic Peptide Levels in Persistent Pulmonary Hypertension
Brief Title: N-Terminal Pro-brain Natriuretic Peptide Hormone and Persistent Pulmonary Hypertension
Status: Terminated | Type: Observational
Why Stopped: Interim analysis showed greater variablility in NT-proBNP findings than anticipated.
Sponsor: Christiana Care Health Services (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: CCC 27004
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2009-05

CONDITIONS: Persistent Pulmonary Hypertension of Newborn
Keywords: Persistent Pulmonary Hypertension; N-terminal pro brain natriuretic peptide
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PPHN: Infants with persistent pulmonary hypertension (PPHN)

SUMMARY:
Babies who are suspected of having persistent pulmonary hypertension (PPHN) will be included in this study. PPHN is a condition in which the blood is restricted from flowing to the lungs in a normal way making it hard for babies to breath and placing strain on the heart. This study will observe whether certain hormones that measure stress (N-terminal pro-brain natriuretic peptide) can help determine how well a baby will do when they have PPHN.

DETAILED DESCRIPTION:
PPHN occurs in infant > or = 34 weeks gestation and is characterized by an elevation in pulmonary vascular resistance (PVR) and right-to-left shunting of the blood at the atrial, ductal, and pulmonary levels, leading to hypoxemia. Management of these infants is complex (and the clinical course) is often difficult to predict.

Brain natriuretic peptide (BNP) is a cardiac hormone that is secreted from cardiac myocytes and cardiac fibroblasts. Upon activation, the prohormone is cleaved into a biologically active BNP and an inactive N-terminal proBNP (NT-proBNP). BNP and NT-proBNP levels are increasingly being used for diagnostic purpose in adults and have been correlated to adult pulmonary hypertension. Multiples studies have been performed to determine normal values for NT-proBNP in the pediatric population. One study measured NT-proBNP levels in umbilical cord blood during the second trimester and at delivery of uncomplicated pregnancies and determined normal reference values of NT-proBNP. It is thought that NT-proBNP has potential for use in term infants with PPHN.

The objective of this research is to correlate NT-proBNP levels to left ventricular dysfunction in term infants with PPHN. Secondarily, we want to assess the possible use of NT-proBNP to predict response to inhaled nitric oxide and the ability to successfully wean off inhaled nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* >/= 34 weeks gestation at birth
* clinical diagnosis of PPHN

Exclusion Criteria:

* newborns with evidence of structural heart disease, congenital anomalies and prior use of inhaled nitric oxide.

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants who are admitted to the NICU with a diagnoses of PPHN.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Euming Chong, MD, Principal Investigator — Christiana Hospital / Thomas Jefferson University Hospital; Constance Andrejko, DO, Principal Investigator — Christiana Hospital / Thomas Jefferson University Hospital
Locations (2):
- United States (2):
  - Christiana Hospital, Newark, Delaware
  - Thomas Jefferson University, Philadelphia, Pennsylvania